CLINICAL TRIAL: NCT01696877
Title: A Neoadjuvant Immunologic Study of Androgen Deprivation Therapy Combined With a Granulocytemacrophage-colony Stimulating Factor F-secreting Allogeneic Prostate Cancer Vaccine and Low-dose Cyclophosphamide in Men With High-risk Localized Prostate Cancer Undergoing Radical Prostatectomy
Brief Title: A Neoadjuvant Study of Androgen Ablation Combined With Cyclophosphamide and GVAX Vaccine for Localized Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: David H. Koch Charitable Foundation (Unknown); BioSante Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1265; NA_00073453 (Other: JHMIRB)
Record Dates: First submitted 2012-09-14; First posted 2012-10-01 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer Adenocarcinoma in Situ
MeSH Terms: interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Degarelix (Active Comparator): Degarelix will be administered as three 80 mg subcutaneous injections, for a total dose of 240 mg at 14 (±3) days prior to surgery. A telephone follow-up interview (or an in-person clinic visit) to evaluate for adverse events will occur 28 (±21) days after prostatectomy. Patients will then be followed by their urologists according to standard institutional practices, but will require prostate-specific antigen evaluations every 3 (±1) months during year 1 and every 6 (±2) months during years 2-3.
  Interventions: Drug: degarelix acetate
- Cyclophosphamide, GVAX and Degarelix (Experimental): Cyclophosphamide will be given at a dose of 200 mg/m2 as a single intravenous infusion. 1 day later, prostate GVAX will be administered as five 0.8-mL intradermal injections of PC3 (2.5 × 108 cells) and five 0.5-mL intradermal injections of LNCaP (2.5 × 108 cells), for a total dose of 5 × 108 cells. On day 14, Degarelix will be administered as three 80 mg subcutaneous injections, for a total dose of 240 mg.
  Interventions: Drug: degarelix acetate; Drug: Cyclophosphamide; Drug: GVAX

INTERVENTIONS:
Drug: degarelix acetate — Degarelix Acetate is a gonadotropin-releasing hormone (GnRH) receptor antagonist. It works by decreasing the amount of testosterone in the body,which the tumor needs to grow.
  Other Names: Firmagon
Drug: Cyclophosphamide — Cyclophosphamide as a potent enhancer of immune responses to GVAX. cyclophosphamide is used as an immune suppressor in many autoimmune disorders.
  Other Names: Cytoxan; Neosar
  Arms: Cyclophosphamide, GVAX and Degarelix
Drug: GVAX — GVAX is granulocytemacrophage -colony stimulating factor -secreting allogeneic cell-based vaccine as immunotherapy for prostate cancer
  Other Names: granulocytemacrophage -colony stimulating factor -secreting cell-based (PC3/LNCaP)immunotherapy
  Arms: Cyclophosphamide, GVAX and Degarelix

SUMMARY:
This research is being done to see if an investigational prostate cancer vaccine, called GVAX, can safely be given together with a single intravenous injection of a drug called cyclophosphamide to men that will undergo surgery to remove their cancerous prostate glands who have also received standard hormonal therapy.

DETAILED DESCRIPTION:
Cancer immunotherapy refers broadly to approaches which attempt to treat cancer by activating immune responses directed against malignant tissue. Prostate GVAX is an allogeneic cell-based prostate cancer vaccine composed of two irradiated cell lines (PC3 and LNCaP) that have been genetically modified to secrete granulocyte-macrophage colony-stimulating factor (granulocytemacrophage-colony stimulating factor). The release of granulocytemacrophage-colony stimulating factor by these modified tumor cells serves to recruit dendritic cells which then present tumor antigens to T-cells, thus initiating antitumor immune responses.

However, abundant preclinical data show that, when used alone, cell-based immunotherapy is unable to break specific T-cell tolerance in tumor-bearing hosts. Studies in an autochthonous prostate cancer mouse model have shown that giving low-dose cyclophosphamide prior to a cell-based granulocytemacrophage-colony stimulating factor-secreting vaccine abrogates immune tolerance through augmentation of CD8+ T cell infiltration in the prostate, transient depletion of regulatory T cells (Tregs), and increased expression of dendritic cell maturation markers. Enhancement of antitumor immunity has also been observed in other preclinical models where cyclophosphamide was given in sequence with granulocytemacrophage-colony stimulating factor-secreting immunotherapy for the treatment of breast and pancreatic cancers. These preclinical data are supported by early-phase clinical trials combining GVAX with low-dose cyclophosphamide in pancreatic and breast cancers.

Furthermore, emerging evidence suggests that androgen deprivation therapy (ADT) itself has profound effects on the host immune system, resulting in thymic regeneration and enhancement of antitumor immunity. In addition, preclinical and clinical studies demonstrate that ADT augments prostate cancer-specific immune responses induced by immunotherapy, suggesting that ADT may act synergistically with immunotherapy. Based on data from mouse models as well as human clinical trials, it has been suggested that prostate cancer immunotherapy may be most effective when administered in the setting of an androgen-suppressed environment.

Building on these findings, investigators have designed a study to assess the use of ADT given alone or administered following immunization with low-dose cyclophosphamide and prostate GVAX, in patients undergoing radical prostatectomy. Investigators aim (1) to determine whether ADT is immunogenic in men with localized prostate cancer by evaluating T-cell infiltration in harvested prostate glands; (2) to determine whether administering ADT after low-dose cyclophosphamide and prostate GVAX augments immune infiltration into the prostate gland; and (3) to investigate whether this combinatorial immuno-hormonal approach is safe and feasible. Investigators hypothesize that the combination of ADT and cyclophosphamide/GVAX will produce significantly greater antitumor immune responses than would ADT used alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate (clinical stage T1c-T3b, N0, M0) without involvement of lymph nodes, bone, or visceral organs
* Initial prostate biopsy is available for central pathologic review, and is confirmed to show at least 2 positive cores and a maximum Gleason sum of ≥ 7
* Radical prostatectomy has been scheduled at Johns Hopkins Hospital
* Age ≥ 21 years
* Eastern Cooperative Oncology Group performance status 0-1, or Karnofsky score ≥ 70%
* Adequate bone marrow, hepatic, and renal function:

  * White Blood Count > 3,000 cells/mm3
  * Absolute neutrophil count > 1,500 cells/mm3
  * Hemoglobin > 9.0 g/dL
  * Platelet count > 100,000 cells/mm3
  * Serum creatinine < 2.0 mg/dL
  * Serum bilirubin < 2 mg/dL
  * Alanine aminotransferase < 2 × upper limit of normal (ULN)
  * Aspartate aminotransferase < 2 × ULN
  * Alkaline phosphatase < 2 × ULN
* Willingness to provide written informed consent and HIPAA authorization for the release of personal health information, and the ability to comply with the study requirements (note: HIPAA authorization will be included in the informed consent)
* Willingness to use barrier contraception from the time of cyclophosphamide and/or GVAX administration until the time of prostatectomy.

Exclusion Criteria:

* Presence of known lymph node involvement or distant metastases
* Other histologic types of prostate cancers such as ductal, sarcomatous, lymphoma, small cell, and neuroendocrine tumors
* Prior radiation therapy, hormonal therapy, biologic therapy, or chemotherapy for prostate cancer
* Prior immunotherapy/vaccine therapy for prostate cancer
* Previous or concurrent use of cyclophosphamide
* Concomitant treatment with other hormonal therapy or 5a-reductase inhibitors
* Current use of systemic corticosteroids or use of corticosteroids within 4 weeks of enrollment (inhaled corticosteroids for asthma or Chronic obstructive pulmonary disease are permitted)
* Use of experimental agents for prostate cancer within the past 3 months
* Known allergy to cyclophosphamide or G-colony stimulating factor /granulocytemacrophage-colony stimulating factor
* Known hypersensitivity to materials of bovine origin (e.g. fetal bovine serum), or other components of GVAX which include Dimethyl sulfoxide and hydroxyethyl starch as well as small amounts of porcine trypsin and DNase
* History or presence of autoimmune disease requiring systemic immunosuppression (including but not limited to: inflammatory bowel disease, systemic lupus erythematosus, vasculitis, rheumatoid arthritis, scleroderma, multiple sclerosis, hemolytic anemia, Sjögren syndrome, and sarcoidosis)
* Other concurrent malignancies, with the exception of non-melanoma skin cancers and superficial bladder cancer
* Uncontrolled major active infectious, cardiovascular, pulmonary, hematologic, or psychiatric illnesses that would make the patient a poor study candidate
* Known prior or current history of HIV and/or hepatitis B/C

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-01-18 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanual Antonarakis, M.D, Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclophosphamide, GVAX and Degarelix: Cyclophosphamide will be given at a dose of 200 mg/m2 as a single intravenous infusion. 1 day later, prostate GVAX will be administered as five 0.8-mL intradermal injections of PC3 (2.5 × 108 cells) and five 0.5-mL intradermal injections of LNCaP (2.5 × 108 cells), for a total dose of 5 × 108 cells. On day 14, Degarelix will be administered as three 80 mg subcutaneous injections, for a total dose of 240 mg.
  degarelix acetate: Degarelix Acetate is a gonadotropin-releasing hormone (GnRH) receptor antagonist. It works by decreasing the amount of testosterone in the body,which the tumor needs to grow.
  Cyclophosphamide: Cyclophosphamide as a potent enhancer of immune responses to GVAX. cyclophosphamide is used as an immune suppressor in many autoimmune disorders.
  GVAX: GVAX is granulocytemacrophage-colony stimulating factor -secreting allogeneic cell-based vaccine as immunotherapy for prostate cancer
Period: Overall Study
Arm/Group | Degarelix | Cyclophosphamide, GVAX and Degarelix
Started | 15 | 14
Completed | 15 | 13
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only participants who were randomized and underwent prostatectomy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix | Cyclophosphamide, GVAX and Degarelix | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 14 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 15 | 12 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Intraprostatic CD8+ T Cell Infiltration
Description: CD8+ T cell infiltration (quantified as log[CD8 density]) into the prostate from harvested prostate glands in men with localized prostate cancer receiving neoadjuvant Androgen deprivation therapy alone (2 weeks prior to surgery), or cyclophosphamide and GVAX followed by Androgen deprivation therapy, (with cyclophosphamide/GVAX administered 4 weeks prior to prostatectomy, and Androgen deprivation therapy administered 2 weeks prior to prostatectomy).
Time Frame: 2 years
Measure: Mean (95% Confidence Interval); unit: log10 (cells/mm^2)
Arm/Group | Degarelix | Cyclophosphamide, GVAX and Degarelix
Number analyzed (Participants) | 15 | 13
log10 (cells/mm^2) | 204.81 [120.67 to 288.95] | 263.33 [129.4 to 397.25]

2. Secondary Outcome: Intraprostatic CD4+ T Cell and Treg Infiltration
Description: Number of participants with CD4+ T cell and Treg infiltration into the prostate.
Time Frame: 2 years
Population: Data was not collected for this outcome measure
Arm/Group | Degarelix | Cyclophosphamide, GVAX and Degarelix
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quantification of Tissue Androgen Concentrations
Description: Tissue androgen concentrations (testosterone, dihydrotestosterone), and androgen receptor (AR) protein expression in prostate specimens
Time Frame: 2 years
Population: Data was not collected for this outcome measure
Arm/Group | Degarelix | Cyclophosphamide, GVAX and Degarelix
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Quantification of Markers of Apoptosis
Description: Amount of apoptosis (activated caspase 3) and proliferation (Ki-67) in prostate tumor specimens
Time Frame: 2 years
Population: Data was not collected for this outcome measure
Arm/Group | Degarelix | Cyclophosphamide, GVAX and Degarelix
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pathological Complete Responses
Description: Number of participants with pathological complete response (pCR)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Cyclophosphamide, GVAX and Degarelix: Cyclophosphamide will be given at a dose of 200 mg/m2 as a single intravenous infusion. 1 day later, prostate GVAX will be administered as five 0.8-mL intradermal injections of PC3 (2.5 × 108 cells) and five 0.5-mL intradermal injections of LNCaP (2.5 × 108 cells), for a total dose of 5 × 108 cells. On day 14, Degarelix will be administered as three 80 mg subcutaneous injections, for a total dose of 240 mg.
  degarelix acetate: Degarelix Acetate is a gonadotropin-releasing hormone (GnRH) receptor antagonist. It works by decreasing the amount of testosterone in the body,which the tumor needs to grow.
  Cyclophosphamide: Cyclophosphamide as a potent enhancer of immune responses to GVAX. cyclophosphamide is used as an immune suppressor in many autoimmune disorders.
  GVAX: GVAX is Granulocyte-macrophage-colony stimulating factor-secreting allogeneic cell-based vaccine as immunotherapy for prostate cancer
Arm/Group | Degarelix | Cyclophosphamide, GVAX and Degarelix
Number analyzed (Participants) | 15 | 13
Participants | 0 | 0

6. Secondary Outcome: Serum Antibodies to Prostate-associated Antigens
Description: Number of participants with generation of novel antibodies to prostate-associated antigens in the serum of patients, after the initiation of protocol therapy
Time Frame: 2 years
Population: Data was not collected for this outcome measure
Arm/Group | Degarelix | Cyclophosphamide, GVAX and Degarelix
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Prostate-specific Antigen Response Rate
Description: Number of participants with Prostate-specific antigen response
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Degarelix | Cyclophosphamide, GVAX and Degarelix
Number analyzed (Participants) | 15 | 13
Participants | 13 | 11

8. Secondary Outcome: Percentage of Participants Without Prostate Specific Antigen Recurrence at 24 Months After Surgery
Description: Percentage of participants in each arm who were free of prostate specific antigen recurrence (i.e. prostate specific antigen remained undetectable after prostatectomy) at 24 months after undergoing surgery.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Degarelix | Cyclophosphamide, GVAX and Degarelix
Number analyzed (Participants) | 15 | 13
percentage of participants | 38 [19 to 74] | 66 [43 to 100]

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events after receiving study drug and before prostatectomy as well as doing each follow up visit after prostatectomy up to 3 years.
Description: An adverse event (AE) is defined as any untoward medical occurrence (symptom, sign, illness or experience) that develops or worsens in a research patient during a clinical study or within 30 days post-treatment, regardless of causality.
Groups:
- Cyclophosphamide, GVAX and Degarelix: Cyclophosphamide will be given at a dose of 200 mg/m2 as a single intravenous infusion. 1 day later, prostate GVAX will be administered as five 0.8-mL intradermal injections of PC3 (2.5 × 108 cells) and five 0.5-mL intradermal injections of LNCaP (2.5 × 108 cells), for a total dose of 5 × 108 cells. On day 14, Degarelix will be administered as three 80 mg subcutaneous injections, for a total dose of 240 mg.
  degarelix acetate: Degarelix Acetate is a gonadotropin-releasing hormone (GnRH) receptor antagonist. It works by decreasing the amount of testosterone in the body,which the tumor needs to grow.
  Cyclophosphamide: Cyclophosphamide as a potent enhancer of immune responses to GVAX. cyclophosphamide is used as an immune suppressor in many autoimmune disorders.
  GVAX: GVAX is GM-CSF-secreting allogeneic cell-based vaccine as immunotherapy for prostate cancer
Arm/Group | Degarelix | Cyclophosphamide, GVAX and Degarelix
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/15 | 2/14
Other Adverse Events (participants affected / at risk) | 15/15 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix (N=15) | Cyclophosphamide, GVAX and Degarelix (N=14)
Hematoma (Vascular disorders) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) — Pulmonary embolism
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix (N=15) | Cyclophosphamide, GVAX and Degarelix (N=14)
Fatigue (General disorders) | 4 (4) | 3 (3)
Injection site reaction (General disorders) | 8 (22) | 12 (50) — erythema bilateral legs
Urinary Incontinence (Renal and urinary disorders) | 4 (4) | 10 (11)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alkaline Phosphatase (Investigations) | 1 (1) | 0 (0) — Increased Alkaline Phosphatase
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Shingles (right side of body)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Premature menopause (Reproductive system and breast disorders) | 7 (7) | 8 (8) — hot flashes
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 2 (3) — nocturia
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 7 (8)
Allergic reaction (Immune system disorders) | 1 (1) | 6 (15) — allergic reaction/erythema
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) — facial nerve disorder (Bell's Palsy)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — nasal congestion
Fever (General disorders) | 0 (0) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) — muscle soreness (legs)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) — lower abdominal pain
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (6)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) — restless/ anxious
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (3) — peri-oral numbness
Weight gain (Investigations) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) — pulmonary embolism
Chills (General disorders) | 1 (1) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) — swollen tongue
Eye disorders - Other, (Eye disorders) | 0 (0) | 1 (1) — soreness around eyes
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT01696877/Prot_SAP_000.pdf